CLINICAL TRIAL: NCT02267317
Title: Phase 2 Study of The Role of Pharmacologic Inhibition of TLR4 With E5564 on Glucose Metabolism in Insulin Resistant Subjects.
Brief Title: The Effect of TLR4 Inhibition in Obese and Type 2 Diabetic Subjects
Acronym: Eritoran2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study drug expired
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC20140498H
Record Dates: First submitted 2014-09-26; First posted 2014-10-17 (Estimated); Results first posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2018-09

CONDITIONS: Insulin Sensitivity
Keywords: Insulin signaling and glucose disposal in muscle; Hepatic insulin sensitivity; TLR4 signaling and inflammatory gene expression; Plasma cytokine concentration; Intramyocellular diacylglycerol and ceramide content
MeSH Terms: conditions — Insulin Resistance | interventions — eritoran; E5564

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Obese Group-D5W (Active Comparator): Obese subjects receive IV administration of 5% Dextrose in water/D5W (vehicle) 12 mg every 12 hours
  Interventions: Drug: D5W
- Obese Group - Eritoran (Active Comparator): Obese subjects receive IV administration of Eritoran 12 mg every 12 hours
  Interventions: Drug: Eritoran
- Diabetes (T2DM) Group - D5W (Active Comparator): T2DM subjects receive IV administration of 5% Dextrose in water/D5W (vehicle) 12 mg every 12 hours
  Interventions: Drug: D5W
- Diabetes (T2DM) Group - Eritoran (Active Comparator): T2DM subjects receive IV administration of Eritoran 12 mg every 12 hours
  Interventions: Drug: Eritoran

INTERVENTIONS:
Drug: Eritoran — Pharmacologic inhibitor of TLR4 receptors.
  Other Names: E5564
  Arms: Diabetes (T2DM) Group - Eritoran; Obese Group - Eritoran
Drug: D5W — 5% Dextrose Water = Vehicle
  Other Names: Placebo, Vehicle
  Arms: Diabetes (T2DM) Group - D5W; Obese Group-D5W

SUMMARY:
To determine whether pharmacologic inhibition of Toll-like receptor 4 (TLR4) with eritoran for injection (E5564) will reduce inflammation and improve glucose metabolism in insulin resistant (obese and T2DM) subjects.

DETAILED DESCRIPTION:
E5564 = Eritoran

ELIGIBILITY:
Inclusion Criteria:

* Subjects capable of giving informed consent.
* lean (BMI <26 kg/m2) with normal glucose-tolerant subjects without a family history of type 2 DM
* obese (BMI 30-37 kg/m2) with normal glucose-tolerant subjects
* Type 2 DM subjects base on ADA criteria, who have HbA1c <8.5% and control with diet or sulfonylureas.
* Both genders. (50% males)
* Age = 18-65 years. Older subjects are excluded because aging is a pro-inflammatory state.
* All ethnic groups
* Premenopausal women in the follicular phase, non-lactating, and with a negative pregnancy test. Postmenopausal women on stable dose of or not exposed to hormone replacement for >=6 months.
* Lab: Hematocrit >=34%, serum creatinine <=1.4 mg/dL, normal electrolytes, urinalysis, and coagulation tests. Liver function tests up to 2x normal range.
* Stable body weight (+/-1%) for >=3 months.
* One or less sessions of strenuous exercise/wk for last 6 months.

Exclusion Criteria:

* Current treatment with drugs known to affect glucose and lipid homeostasis. Subjects on a stable dose of statin (>3 months) are eligible.
* Non-steroidal anti-inflammatory drugs or systemic steroid use for more than 1 week within 3 months.
* Current treatment with anticoagulants (warfarin). Aspirin (up to 325 mg) and clopidogrel will be permitted if these can be held for seven days prior to the biopsies.
* History of heart disease (New York Heart Classification greater than class II; more than non-specific ST-T wave changes on the ECG), peripheral vascular disease, pulmonary disease, smokers.
* Poorly controlled blood pressure (systolic BP>160, diastolic BP>90 mmHg).
* Active inflammatory, autoimmune, infectious, hepatic, gastrointestinal, malignant, and psychiatric disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-01; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Musi, MD, Principal Investigator — Audie L. Murphy VA Hospital, STVHCS San Antonio, Texas, United States 78229
Locations (1):
- Audie L. Murphy VA Hospital, STVHCS, San Antonio, Texas, United States

REFERENCES:
- [Derived] Liang H, Sathavarodom N, Colmenares C, Gelfond J, Espinoza SE, Ganapathy V, Musi N. Effect of acute TLR4 inhibition on insulin resistance in humans. J Clin Invest. 2022 Nov 1;132(21):e162291. doi: 10.1172/JCI162291. PMID 36066991

RESULTS

PARTICIPANT FLOW:
Groups:
- Obese Group - D5W - Eritoran: Obese subjects randomized to receive D5W first, then Eritoran
- Obese Group - Eritoran - D5W: Obese subjects randomized to receive Eritoran first, then D5W.
- Diabetes (T2DM) Group - D5W - Eritoran: T2DM subjects randomized to receive D5W first then Eritoran
- Diabetes (T2DM) Group - Eritoran - D5W: T2DM subjects randomized to receive Eritoran first then D5W
- Lean Group - D5W - Eritoran: Lean subjects randomized to receive D5W first then Eritoran
- Lean Group - Eritoran - D5W: Lean subjects randomized to receive Eritoran first then d5W
Period: Infusion1
Arm/Group | Obese Group - D5W - Eritoran | Obese Group - Eritoran - D5W | Diabetes (T2DM) Group - D5W - Eritoran | Diabetes (T2DM) Group - Eritoran - D5W | Lean Group - D5W - Eritoran | Lean Group - Eritoran - D5W
Started | 8 | 3 | 1 | 2 | 0 | 1
Completed | 8 | 3 | 1 | 2 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (3-4weeks Between Infusions)
Arm/Group | Obese Group - D5W - Eritoran | Obese Group - Eritoran - D5W | Diabetes (T2DM) Group - D5W - Eritoran | Diabetes (T2DM) Group - Eritoran - D5W | Lean Group - D5W - Eritoran | Lean Group - Eritoran - D5W
Started | 8 | 3 | 1 | 2 | 0 | 1
Completed | 6 | 3 | 1 | 2 | 0 | 1
Not Completed | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Period: Infusion2
Arm/Group | Obese Group - D5W - Eritoran | Obese Group - Eritoran - D5W | Diabetes (T2DM) Group - D5W - Eritoran | Diabetes (T2DM) Group - Eritoran - D5W | Lean Group - D5W - Eritoran | Lean Group - Eritoran - D5W
Started | 6 | 3 | 1 | 2 | 0 | 1
Completed | 6 | 3 | 1 | 2 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Obese Group: Subjects with BMI >30 kg/m2 were enrolled to receive two infusions, the order of which was randomly assigned.
- Type 2 Diabetic Subjects: Subjects with BMI >30 kg/m2 and 2-hour Oral Glucose Tolerance Test >200mg/dL
- Lean/Healthy: Subjects with BMI <26 kg/m2 and normal glucose tolerant
- Total: Total of all reporting groups
Arm/Group | Obese Group | Type 2 Diabetic Subjects | Lean/Healthy | Total
Number analyzed (Participants) | 11 | 3 | 1 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (6.0) | 55 (15.6) | 19 (0) | 53 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 0 | 8
  Male | 4 | 2 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 1 | 1 | 11
  Not Hispanic or Latino | 1 | 2 | 0 | 3
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 11 | 3 | 1 | 15
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.1 (1.8) | 33.5 (3.3) | 19 (0) | 31.5 (4.0)
HbA1c [Mean (Standard Deviation); unit: Percentage of glycated hemoglobin] | 5.4 (0.2) | 6.3 (0.7) | 5.3 (0) | 5.6 (0.5)
Fasting plasma glucose [Mean (Standard Deviation); unit: mg/dL] | 5.1 (0.8) | 6.9 (0.7) | 4.5 (0) | 5.4 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Effect of Eritoran on Muscle Insulin Sensitivity
Description: Muscle insulin sensitivity = muscle insulin sensitivity is determined by euglycemic hyperinsulinemic clamp procedure. M value (mg glucose / kg of body weight / minute) calculated from the clamp is measured. Higher M value indicates better insulin sensitivity. There is no established reference range.
Time Frame: 72 hours
Population: Data from T2DM subjects and Lean subject were not collected for primary outcome measure because of insufficient number of participants in the 2 groups.
Measure: Mean (Standard Error); unit: mg/kg/min
Groups:
- Obese Group - Placebo: Obese subjects - IV administration of D5W (5% Dextrose in water)
- Obese Group - Eritoran: Obese subjects - IV administration of Eritoran 12 mg every 12 hours
- Diabetes (T2DM) Group - Placebo: T2DM subjects - IV administration of D5W (5% Dextrose in water)
- Diabetes (T2DM) Group - Eritoran: T2DM subjects - IV administration of Eritoran 12 mg every 12 hours
- Lean - Placebo: Lean subjects - IV administration of D5W (5% Dextrose in water)
- Lean - Eritoran: Lean subjects - IV administration of Eritoran 12 mg every 12 hours
Arm/Group | Obese Group - Placebo | Obese Group - Eritoran | Diabetes (T2DM) Group - Placebo | Diabetes (T2DM) Group - Eritoran | Lean - Placebo | Lean - Eritoran
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0 | 0
mg/kg/min | 8.0 (0.9) | 10.6 (1.1) |  |  |  |

2. Primary Outcome: Effect of Eritoran on Hepatic Insulin Sensitivity
Description: Hepatic insulin sensitivity = is determined by euglycemic hyperinsulinemic clamp procedure. Endogenous glucose production or EGP (mg/kg/min) calculated from the clamp is measured. Lower EGP indicates better hepatic insulin sensitivity. There is no established reference range.
Time Frame: 72 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/kg/min
Arm/Group | Obese Group - Placebo | Obese Group - Eritoran | Diabetes (T2DM) Group - Placebo | Diabetes (T2DM) Group - Eritoran | Lean - Placebo | Lean - Eritoran
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0 | 0
mg/kg/min | 2.0 (0.2) | 1.9 (0.1) |  |  |  |

3. Secondary Outcome: Effect of Eritoran on TLR4 Expression in Muscle Tissue
Description: TLR4 expression in muscle tissue is determined by RNAseq using arbitrary units. Higher TLR4 expression indicates higher inflammatory response. There is no reference range.
Time Frame: 72 hours
Population: The total number of obese subjects enrolled is 9. However, we were only able to obtain muscle biopsies from 7 subjects. In addition, data from T2DM subjects and Lean subject were not collected for this secondary outcome measure because of insufficient number of participants in the 2 groups.
Measure: Mean (Standard Error); unit: AU
Arm/Group | Obese Group - Placebo | Obese Group - Eritoran | Diabetes (T2DM) Group - Placebo | Diabetes (T2DM) Group - Eritoran | Lean - Placebo | Lean - Eritoran
Number analyzed (Participants) | 7 | 7 | 0 | 0 | 0 | 0
AU | 1 (0.11) | 1.16 (0.16) |  |  |  |

4. Secondary Outcome: Effect of Eritoran on TLR4 Expresison in Adipose Tissue
Description: TLR4 expression in the adipose tissue is determined by RNAseq using arbitrary units. Higher TLR4 expression indicates higher inflammatory response. There is no reference range.
Time Frame: 72 hours
Population: The total number of obese subjects enrolled is 9. However, we were only able to obtain fat biopsies from 4 subjects. In addition, data from T2DM subjects and Lean subject were not analyzed for this secondary outcome measure because of insufficient number of participants in the 2 groups.
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Obese Group - Placebo | Obese Group - Eritoran | Diabetes (T2DM) Group - Placebo | Diabetes (T2DM) Group - Eritoran | Lean - Placebo | Lean - Eritoran
Number analyzed (Participants) | 4 | 4 | 0 | 0 | 0 | 0
AU | 1 (0.11) | 1.22 (0.07) |  |  |  |

5. Secondary Outcome: Effect of Eritoran on TLR4 Expression in Peripheral Blood Monocytes
Description: TLR4 expression in the peripheral blood monocytes is determined by flow cytometry using arbitrary units. Higher TLR4 expression indicates higher inflammatory response. There is no reference range.
Time Frame: 72 hours
Population: Data from T2DM subjects and Lean subject were not analyzed because the number of participants was insufficient in the 2 groups.
Measure: Mean (Standard Error); unit: AU
Arm/Group | Obese Group - Placebo | Obese Group - Eritoran | Diabetes (T2DM) Group - Placebo | Diabetes (T2DM) Group - Eritoran | Lean - Placebo | Lean - Eritoran
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0 | 0
AU | 1.1 (0.1) | 1.2 (0.1) |  |  |  |

6. Secondary Outcome: Effect of Eritoran on Plasma TNF-alpha (Tumor Necrosis Factor-alpha) Concentration
Description: TNF-alpha levels are determined by ELISA. Higher level indicates higher inflammatory response. There is no established reference range.
Time Frame: 72 hours
Population: as for outcome 5
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Obese Group - Placebo | Obese Group - Eritoran | Diabetes (T2DM) Group - Placebo | Diabetes (T2DM) Group - Eritoran | Lean - Placebo | Lean - Eritoran
Number analyzed (Participants) | 9 | 9 | 0 | 0 | 0 | 0
pg/ml | 2.4 (0.3) | 2.3 (0.2) |  |  |  |

7. Secondary Outcome: Effect of Eritoran on Intramyocellular Diacylglycerol and Ceramide Content
Description: Intramyocellular diacylglycerol and ceramide content are determined by mass spectrometry. Higher levels have been associated with diabetes.
Time Frame: 72 hours
Population: Data were not collected due to lack of funding.
Arm/Group | Obese Group - Placebo | Obese Group - Eritoran | Diabetes (T2DM) Group - Placebo | Diabetes (T2DM) Group - Eritoran | Lean - Placebo | Lean - Eritoran
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 19 months
Groups:
- Lean/Healthy Group - Placebo: Lean subjects - IV administration of D5W (5% Dextrose in water)
- Lean/Healthy Group - Eritoran: Lean subjects - IV administration of Eritoran 12 mg every 12 hours
Arm/Group | Obese Group - Placebo | Obese Group - Eritoran | Diabetes (T2DM) Group - Placebo | Diabetes (T2DM) Group - Eritoran | Lean/Healthy Group - Placebo | Lean/Healthy Group - Eritoran
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/3 | 0/3 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/3 | 0/3 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 9/11 | 9/11 | 1/3 | 2/3 | 0/1 | 0/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Obese Group - Placebo (N=11) | Obese Group - Eritoran (N=11) | Diabetes (T2DM) Group - Placebo (N=3) | Diabetes (T2DM) Group - Eritoran (N=3) | Lean/Healthy Group - Placebo (N=1) | Lean/Healthy Group - Eritoran (N=1)
Phlebitis Grade 1, 2 or 3 (Vascular disorders) | 7 | 9 | 1 | 2 | 0 | 0
Dermatology (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hot flashes (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypokalemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 3 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT02267317/Prot_SAP_000.pdf